CLINICAL TRIAL: NCT01333891
Title: Choroidal Thickness During Changes in Intraocular Pressure and Arterial Blood Pressure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv. Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OPHT-151010
Record Dates: First submitted 2011-04-11; First posted 2011-04-12 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
MeSH Terms: interventions — Phenylephrine; Nitroprusside; Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sodium-Nitroprusside (Active Comparator): Nipruss®, Sanol-Schwarz, Monheim, Germany 0, 0.5, 1 and 2 µg/kg/min, each infusion step for 5 minutes, total infusion period of 20 minutes
  Interventions: Drug: Phenylephrine; Drug: Sodium-Nitroprusside; Device: Suction Cup; Device: Goldmann applanation tonometer; Device: 1060nm Optical coherence tomography
- Phenylephrine (Active Comparator): Neosynephrine®, Winthrop Breon Laboratories New York, NY, USA 0, 0.5, 1 and 2 μg/kg/min, each infusion step for 5 minutes, total infusion period of 20 minutes
  Interventions: Drug: Phenylephrine; Drug: Sodium-Nitroprusside; Device: Suction Cup; Device: Goldmann applanation tonometer; Device: 1060nm Optical coherence tomography
- Suction Cup (Active Comparator): suction force of 25, 50, 75, and 100 mmHg
  Interventions: Drug: Phenylephrine; Drug: Sodium-Nitroprusside; Device: Suction Cup; Device: Goldmann applanation tonometer; Device: 1060nm Optical coherence tomography

INTERVENTIONS:
Drug: Phenylephrine — Neosynephrine®, Winthrop Breon Laboratories New York, NY, USA 0, 0.5, 1 and 2 μg/kg/min, each infusion step for 5 minutes, total infusion period of 20 minutes
Drug: Sodium-Nitroprusside — Nipruss®, Sanol-Schwarz, Monheim, Germany 0, 0.5, 1 and 2 µg/kg/min, each infusion step for 5 minutes, total infusion period of 20 minutes
Device: Suction Cup — experimental stepwise increase of intraocular pressure while measurement of choroidal thickness suction force of 25, 50, 75, and 100 mmH
Device: Goldmann applanation tonometer — intraocular pressure measurements
Device: 1060nm Optical coherence tomography — Optical coherence tomography is a widely used non-invasive method to image the retina and choroid. Using a 1060nm light source coupled to a commercially available OCT system (Heidelberg Engineering, Heidelberg, Germany) allows for the measurement of choroidal thickness

SUMMARY:
Age-related macular degeneration (AMD) and glaucoma are among the leading causes of blindness in the western world. Elevated intraocular pressure (IOP) is a well known major risk factor for glaucoma. In addition, there is growing evidence that vascular factors, including arterial hypertension and hypotension, may play a role in the pathogenesis of AMD and glaucoma. To gain more insight into these mechanisms in humans is the primary goal of the present study.

Optical coherence tomography (OCT) delivers three dimensional, volumetric reflectivity information through transparent media in vivo. Moreover, the images show a high choroidal penetration and a resolution comparable to an histologic examination when infrared light sources are used. Because of its non-invasive character, OCT provides an ideal method for diagnosis and monitoring of retinal and choroidal abnormalities.

The present study aims to investigate whether choroidal thickness is temporarily altered by changes in IOP or systemic hemodynamic parameters. IOP will be increased by the use of a suction cup technique, mean arterial blood pressure will be altered by intravenously administered Phenylephrine or Sodium-Nitroprusside.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years, nonsmokers
* Men and women will be included in equal parts
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal findings in the laboratory testings unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia less than 1 diopter

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug (except oral contraceptives)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks History of hypersensitivity to the trial drugs or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* History of migraine
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2012-12; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Choroidal thickness | 18 months

SECONDARY OUTCOMES:
Systolic/diastolic blood pressure (non-invasive) | 18 months
Intraocular pressure (IOP) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, MD, PD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria